CLINICAL TRIAL: NCT05172713
Title: Outcomes of Patients Who Had an Incomplete Colonoscopy After a Positive Fecal Immunological Test: Study of Practices in the Grand-Est
Brief Title: Outcomes of Patients Who Had an Incomplete Colonoscopy After a Positive Fecal Immunological Test
Acronym: ColonoScopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8090
Record Dates: First submitted 2021-10-13; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Immunological test; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, colorectal cancer (CRC) is the second leading cause of cancer death. Its organized screening (Organized ColoRectal Cancer Screening: DOCCR), now carried out by immunological test for occult blood in the stool, has proven its effectiveness. When the immunological test is positive, the Haute Autorité de Santé recommends a total colonoscopy. In 5 to 10% of cases, this colonoscopy is incomplete. The renewal of the endoscopic procedure or the performance of additional second-line examinations are then recommended. At present, however, the respective place of second-line examinations to be performed in this situation is not the subject of specific and validated recommendations.

ELIGIBILITY:
Inclusion criteria:

* Age between 50 and 75 years old at the time of the colonoscopy
* With incomplete colonoscopy performed in 2018 after a positive fecal immunological test as part of the DOCCR
* Patient whose follow-up has ended
* Patient living in the Grand-Est region and in the department of the site concerned
* Examination carried out by a gastroenterologist from the Grand-Est region
* Subject not having expressed, after information, his opposition to the reuse of his data for the purposes of this research

Exclusion criteria:

* Age ≥ 76 years at the time of colonoscopy
* Colonoscopy performed after a positive Hemoccult® test (screening technique older than the immunological test and different sensitivity / specificity)
* Colonoscopy performed before the fecal immunological test
* Gastroenterologist performing the examination practicing outside the Grand-Est region
* Subject not able to understand the objectives of this research
* Subject under judicial control
* Subject under tutorship or curatorship

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject aged between 50 and 75 years old at the time of the colonoscopy with incomplete colonoscopy performed in 2018 after a positive fecal immunological test as part of the DOCCR
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-16 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04-16 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the patient outcomes who had an incomplete colonoscopy after a positive immunological fecal test | Files analysed retrospectively from January 01, 2018 to December 31, 2018 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service Hépato-Gastroentérologie et Assistance Nutritive - Hôpitaux Universitaires de Strasbourg, Strasbourg, France